CLINICAL TRIAL: NCT04896723
Title: Sexual Dysfunction in Patients With Chronic Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 272717
Record Dates: First submitted 2021-05-05; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Liver Diseases; Liver Cirrhosis
MeSH Terms: conditions — Liver Diseases; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic liver disease
  Interventions: Diagnostic Test: Sexual function questionnaire
- Healthy volunteers
  Interventions: Diagnostic Test: Sexual function questionnaire

INTERVENTIONS:
Diagnostic Test: Sexual function questionnaire — Sexual function questionnaire and cognitive screening assessments

SUMMARY:
This project will determine the incidence of sexual dysfunction in patients with chronic liver disease, through questionnaires. The questionnaires have been designed to assess several facets of sexual health, e.g. libido, physical symptoms, depression, etc. 150 patients in our liver outpatient department, and 150 healthy volunteers will be asked to fill in the questionnaire in paper form. The results of this project will be used to produce patient resources, advice sheets and educational materials for patients with chronic liver disease. There is also scope to consider possible interventions in the future to improve sexual dysfunction in patients with chronic liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a chronic liver disease (including those who have had liver transplantation)
* Aged 18-75
* Able to give informed written consent

Exclusion Criteria:

* Major psychiatric disease
* Patients who lack capacity
* Patient with no chronic liver disease
* Patients not proficient in English

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with chronic liver disease
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with sexual dysfunction | 12 months
  The number of patients suffering from sexual dysfunction in patients with chronic liver disease

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver Studies, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No